CLINICAL TRIAL: NCT02499458
Title: Prospective Validation of Circulating Tumor Cells (CTCs) and Circulating Endothelial Cells (CECs) as Prognostic Biomarkers in Clear Cell Renal Cancer
Brief Title: Prospective Validation of Circulating Tumor Cells & Circulating Endothelial Cells as Biomarkers in Renal Cancer
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Alison Allan, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 105484
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Clear Cell Renal Cancer; Circulating Tumor Cells; Circulating Endothelial Cells; Prognostic Biomarkers; Predictive Biomarkers
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: None- observational study

SUMMARY:
Circulating tumor cells (CTCs) have prognostic value in several tumor types, and increasing evidence suggests that molecular characterization of CTCs can serve as a "liquid biopsy" to understand and address treatment resistance. The goal of this proposal is to demonstrate that CTCs can be accurately enumerated and characterized in metastatic clear cell renal cancer (CCRC) and can serve as prognostic/predictive biomarkers to improve treatment. The challenge surrounding CTC analysis in CCRC is that most CTC technologies (including the clinical gold-standard CellSearch®) depend in epithelial markers such as EpCAM that are expressed at low or heterogeneous levels in CCRC. Members of the research team have developed a novel CTC microfluidic technology that can effectively detect CTCs that are completely undetectable by CellSearch® because of very low EpCAM expression, as well as allowing for CTC recovery for downstream molecular characterization. The goal of this proposal is therefore to test the hypotheses that (1) The microfluidics CTC technology will have better sensitivity/specificity relative to the CellSearch in metastatic CCRC; and (2) Enumeration of CTCs in metastatic CCRC patients (n=66) will have prognostic value, while molecular characterization of CTCs for expression of biomarkers (VHL, VEGF, mTOR, HIF1/HIF2, AKT) related to CCRC etiology will be predictive of response/resistance to targeted therapies. Although CCRC is relatively uncommon, the lack of established adjuvant treatments and high cost of targeted therapies in the palliative setting makes the search for new prognostic/predictive biomarkers an important clinical goal.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status 0-2
2. Age over 18 years
3. Diagnosed renal cancer with clear cell histology
4. Metastatic disease
5. Predicted life expectancy over 2 months
6. Targeted treatment with an anti-VEGF or anti-mTOR agent as first or second line therapy
7. Standard imaging evaluation 4 weeks prior to inclusion
8. Planned for standard imaging within 16 weeks after start of therapy

Exclusion Criteria:

1. Presence of substantial comorbidities (uncontrolled heart or respiratory dysfunction, severe renal or hepatic impairment [Cl Cr below 30ml/h OR Bb>3X ULN])
2. History of a malignancy other than non-melanoma skin cancer in the previous 5 years
3. Any other contraindication to targeted treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology care centre
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity/specificity of CTC enumeration (microfluidics vs CellSearch) | 24 months
  For comparison of the 2 CTC platforms, a Bland-Altman plot will be constructed. This plot is superior to standard correlation statistics in that it assesses agreement rather than association. Initially we will use a Chi-Square test to compare the 2 methods at a cutoff point of ≥5 versus <5 CTCs/7.5mL, with simple comparison of PFS at this level. As the cut-off point may not be the same for each method, we will also compare the methods using simple 2X2 contingency tables.
Progression free survival (PFS). | 24 months
  Survival analysis will be performed by Kaplan Meier and significance analysis will use the log-rank test. Cox multivariate analysis will be performed to look at the number and molecular characteristics of CTCs as independent prognostic parameters of survival.

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  Survival analysis will be performed by Kaplan Meier and significance analysis will use the log-rank test. Cox multivariate analysis will be performed to look at the number and molecular characteristics of CTCs as independent prognostic parameters of survival.
Radiological response | within 16 weeks after start of study
  Radiological assessment of disease status will be carried out as standard-of-care and subjected to correlative analysis relative to CTC status, PFS and OS.
Molecular characterization of CTCs | baseline, 4-6 weeks after start of therapy, 10-12 weeks after start of therapy, post-progression (up to 24 months)
  CTCs will be recovered from the microfluidics device and subjected to molecular characterization for expression of markers related to angiogenesis and hypoxia.
Enumeration of CECs | baseline, 4-6 weeks after start of therapy, 10-12 weeks after start of therapy, post-progression (up to 24 months)
  CTCs will be enumerated on both the CellSearch and the novel microfluidic device.

CONTACTS AND LOCATIONS:
Overall Officials: Alison L Allan, PhD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada